CLINICAL TRIAL: NCT05664581
Title: A Single-Center, Prospective Study to Evaluate the Safety and Effectiveness of Multi-Treatment Regimen With Zeltiq Aesthetics, Inc. Rapid Acoustic Pulse (RAP)™ Device for the Improvement in the Appearance of Cellulite
Brief Title: A Study to Assess the Adverse Events and Effectiveness of Rapid Acoustic Pulse (RAP) Device for the Appearance of Cellulite in Adult Participants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-06
Record Dates: First submitted 2022-12-15; First posted 2022-12-23 (Actual); Results first posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Cellulite
Keywords: Rapid Acoustic Pulse; RAP; Cellulite
MeSH Terms: conditions — Cellulite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Rapid Acoustic Pulse (RAP) (Experimental): Participants will receive 3 separate RAP cellulite treatments sessions.
  Interventions: Device: Rapid Acoustic Pulse

INTERVENTIONS:
Device: Rapid Acoustic Pulse — Transdermal Rapid Acoustic Pulse Treatments

SUMMARY:
Cellulite is the rippling or dimpling of the skin most commonly located on the thighs and buttocks of women. Its appearance and texture are often likened to that of "cottage cheese" or an orange peel. Rapid Acoustic Pulse (RAP) is an electrohydraulic (EH) device developed to improve the appearance of cellulite through microscopic disruption of the connection between the skin and underlying tissue leading to a reduction in the severity of dimples and ridges. The purpose of this study is to assess adverse events and effectiveness of RAP in adults seeking treatment of cellulite.

RAP is an FDA approved device for the short-term improvement in the appearance of cellulite in the buttocks and thighs. Participants 18-50 years of age seeking treatment of cellulite will be enrolled. Up to 15 participants will be enrolled in the study at 1 site in the United States.

Participants will receive 3 separate cellulite treatment sessions. Each treatment session will consist of RAP treatment delivered to bilateral thigh and/or buttock areas using the same treatment settings for both sides. The study duration is up to 72 weeks.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a clinic. The effect of the treatment will be checked by medical assessments, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participants seeking treatment of cellulite in the thigh and/or buttock areas.
* Areas of moderate to severe cellulite on bilateral thigh and/or buttock using the Cellulite Dimple - At Rest Scale at Baseline with grades of 2 or 3 based on review of photos taken under the same lightening conditions planned for the trial.
* Participant will not have had invasive or energy-based cellulite (liposuction, subcision, RF, laser, ESWT, cryo-lipolysis, muscle stimulation, etc.) treatments in the treatment areas in the prior 12 months.
* Participant will not have used topical based cellulite treatments for prior 3 months and will not use during the trial
* Participant will not have used spray-on tanning treatments for 3 months prior to or during the term of the trial.

Exclusion Criteria:

* Metal or plastic implants (vascular stent, or implants in the hips, knees, etc.) in the treatment areas.
* Active electronic implants such as pacemakers, defibrillators
* History of coagulopathy and/or on anticoagulant medication
* Skin disorders (skin infections or rashes, psoriasis, etc.) in the treatment areas.
* Medical disorder that would hinder wound healing or immune response.
* Any surgical procedure in the treatment areas in the prior 3 months or planned during the duration of the study.
* Any other condition/disease/situation which, as deemed by the PI, would preclude participant from safely participating in or completing the study visits or that may confound study results.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 14 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zeltiq Aesthetics, Study Director — Zeltiq Aesthetics
Locations (1):
- Innovation Research Center, Pleasanton, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fourteen participants were enrolled at 1 study site in the United States.
Pre-assignment Details: The Full Analysis Set (FAS) included all participants who received three assigned treatments with the device and completed the 12-week follow-up visit per the protocol (N=14). The Safety Analysis Set included all enrolled participants who received any treatments (N=14).
Groups:
- All Participants: Participants received 3 separate transdermal Rapid Acoustic Pulse (RAP) cellulite treatment sessions on weeks 1, 4, and 16 delivered to bilateral thigh and/or buttock areas using the same treatment settings for both sides.
Period: Overall Study
Arm/Group | All Participants
Started | 14
Completed | 12
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Safety Population
Arm/Group | All Participants
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.5 (5.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Before and After Side-by-side Photographs Correctly Identified by At Least 2 of 3 Blinded Reviewers From the Independent Physician Reviewer (IPR) Panel
Description: Photographs of the treatment areas were taken at baseline, and at 12-weeks after post-final treatment to determine if the RAP treatment had the effect of improvement in the appearance of cellulite. The photographs were assessed by blinded independent reviewers (IPR) to correctly identify the 12-weeks post-treatment photographs from randomly placed side-by-side comparison of before and after photographs. Reported here is the percentage (%) of images that were correctly identified by at least 2 out of 3 blinded independent reviewers.
Time Frame: Baseline, 12 weeks post-final treatment
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: % of images identified correctly
Units Other Than Participants: Photographs
Arm/Group | All Participants
Number analyzed (Participants) | 14
Number analyzed (Photographs) | 14
% of images identified correctly | 71.4 [41.9 to 91.6]

2. Primary Outcome: Number of Participants With Device-related or Treatment-related: Adverse Events (AEs), Serious AEs (SAEs), Adverse Device Events (ADEs), Serious ADEs (SADEs), Unanticipated AEs or Unanticipated ADEs
Description: An adverse event (AE) was defined as any unfavorable or unintended sign, symptom, or disease that occurred or was reported by the participant to have occurred, or a worsening of a pre-existing condition. A SAE resulted in death, was life threatening, required hospitalization, was a persistent or significant disability/incapacity, a birth defect, or was an event that required medical intervention. An ADE was defined as any AE with a reasonable possibility (definitely, probably, possibly, or remotely related) that the event may have been caused by the study device only.
Time Frame: Week 1 up to 52 weeks post-final treatment
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 14
Participants
  AEs | 2
  SAEs | 0
  ADEs | 2
  SADEs | 0
  Unanticipated AEs | 2
  Unanticipated ADEs | 0

3. Secondary Outcome: Number of Participants With "Agree" or "Strongly Agree" Responses to the Participant Satisfaction Survey in the Improvement in Appearance of Cellulite
Description: The study participant responded to the Participant Satisfaction Survey statement, "In comparison to the pre-treatment photo, the 12 week photograph of the treatment area appears improved." Response choices to this statement were "Strongly Agree", "Agree", "Neutral", "Disagree", and "Strongly Disagree", with "Strongly Agree" representing the greatest perceived improvement in the appearance of cellulite. Reported here is the number of participants who responded with "Agree" or "Strongly Agree." Data are reported for response to photographs on the left and right side of the body.
Time Frame: Baseline, 12 weeks post-final treatment
Population: Full Analysis Set
Measure: Number; unit: participants
Units Other Than Participants: images
Arm/Group | All Participants
Number analyzed (Participants) | 14
Number analyzed (images) | 14
participants | 5

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from first treatment up to 52 weeks post-final treatment.
Groups:
- All Participants: Participants received 3 separate transdermal Rapid Acoustic Pulse (RAP) cellulite treatment sessions on weeks 1, 4, and 16 delivered to bilateral thigh and/or buttock areas using the same treatment settings for both sides, and then were followed for up to 52 weeks post-last treatment.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 2/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=14)
Application Site Discoloration (General disorders) | 2 (2)
Blister (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patentor proprietary protection.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT05664581/Prot_SAP_001.pdf